CLINICAL TRIAL: NCT02508012
Title: Medico-economic Evaluation of the Therapeutic Drug Monitoring of Anti-TNF Agents in the Management of Patients With Inflammatory Bowel Disease Treated With Anti-TNFalpha Biotherapy.
Brief Title: Medico-economic Evaluation of the Therapeutic Drug Monitoring of Anti-TNF-α Agents in Inflammatory Bowel Diseases
Acronym: ATAIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Department of the medical information of Montpellier (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9535
Record Dates: First submitted 2015-07-23; First posted 2015-07-24 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: anti-TNF; Immuno-monitoring; Anti-drug antibody (ADAb); Inflammatory bowel disease (IBD); Crohn's disease; Ulcerative colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immuno monitoring (Experimental): in case of loss of response, the clinician uses immunomonitoring data to adapt the treatment following a treatment algorithm.
  Interventions: Other: Immuno monitoring
- No immuno monitoring (No Intervention): in case of loss of response, immunomonitoring data are not transmit to the clinician who adapts the treatment with classical biological informations.

INTERVENTIONS:
Other: Immuno monitoring — treatment optimization
  Arms: Immuno monitoring

SUMMARY:
Since their appearance more than a decade ago, anti-tumor necrosis factor (TNF) inhibitors have demonstrated beneficial activity in the treatment of inflammatory bowel diseases (IBD). However, more than one-third of patients present primary resistance, and one more third become resistant over time. One of the main factors associated with loss of response is the immunogenicity of anti-TNF biologics leading to the production of antibodies targetting the TNF inhibitor, namely anti-drug antibodies (ADAbs), that accelerate drug elimination from the serum and decrease its therapeutic activity. In this study the investigators propose a medico-economic evaluation of the measurement of anti-TNF agents and anti-drug antibodies serum concentrations in the management of patients with inflammatory bowel disease treated with anti-TNFalpha inhibitors. 280 patients with Crohn's disease (CD) or ulcerative colitis (UC) will be included and randomized in 2 groups with or without drug and ADAbs monitoring. In the monitored group, in case of loss of response, the clinician will use biological informations to adapt the treatment following a simple treatment algorithm. In the unmonitored group, drug and ADAbs measurements will not be transmitted to the clinician. Clinical and economical benefits of the biological monitoring will be evaluated after a follow-up period of two years.

DETAILED DESCRIPTION:
280 patients with Crohn's disease (CD) or ulcerative colitis (UC) will be recruited in 13 french centers and randomized in 2 groups with or without drug and ADAbs monitoring.

Anti-TNF inhibitors and ADAbs will be simultaneously measured in the patients serum by ELISA (LisaTracker - Theradiag) at weeks 6 and 24, months 4, 8, 12, 16, 20 and 24.

In the unmonitored group, drug and ADAbs measurements will not be transmitted to the clinician.

In the monitored group, in case of loss of response the clinician will use immunomonitoring data to adapt the treatment following a simple treatment algorithm:

* loss of response with therapeutic serum trough level of anti-TNF switch to another biologic
* loss of response with subtherapeutic serum trough level of anti-TNF but without detectable ADAbs increase doses and/or shorten interval between infusions
* loss of response with subtherapeutic serum trough level of anti-TNF and detectable ADAbs switch to another anti-TNF if inefficient switch to another biologic.

Clinical and economical benefits of the biological monitoring will be evaluated after a follow-up period of two years:

* primary outcome: Cost-utility analysis of the immunomonitoring strategy using incremental cost effectiveness ratio
* secondary outcome: Evaluation of the quality of life (IBDQ score)

ELIGIBILITY:
Inclusion Criteria:

* patients with Crohn's disease or ulcerative colitis
* Treated with anti-TNF

Exclusion Criteria:

* anti-TNF contraindication
* Previous treatment with anti-TNF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
cost-utility analysis of the immunomonitoring strategy | 2 years
  incremental cost-effectiveness ratio

SECONDARY OUTCOMES:
quality of life | 2 years
  IBDQ score

CONTACTS AND LOCATIONS:
Overall Officials: Thierry VINCENT, MD, PhD, Principal Investigator — Department of immunology in Montpellier
Locations (1):
- University hospital, Montpellier, France

REFERENCES:
- [Background] Baert F, Noman M, Vermeire S, Van Assche G, D' Haens G, Carbonez A, Rutgeerts P. Influence of immunogenicity on the long-term efficacy of infliximab in Crohn's disease. N Engl J Med. 2003 Feb 13;348(7):601-8. doi: 10.1056/NEJMoa020888. PMID 12584368
- [Background] Bartelds GM, Wijbrandts CA, Nurmohamed MT, Stapel S, Lems WF, Aarden L, Dijkmans BA, Tak PP, Wolbink GJ. Clinical response to adalimumab: relationship to anti-adalimumab antibodies and serum adalimumab concentrations in rheumatoid arthritis. Ann Rheum Dis. 2007 Jul;66(7):921-6. doi: 10.1136/ard.2006.065615. Epub 2007 Feb 14. PMID 17301106
- [Background] de Vries MK, Brouwer E, van der Horst-Bruinsma IE, Spoorenberg A, van Denderen JC, Jamnitski A, Nurmohamed MT, Dijkmans BA, Aarden LA, Wolbink GJ. Decreased clinical response to adalimumab in ankylosing spondylitis is associated with antibody formation. Ann Rheum Dis. 2009 Nov;68(11):1787-8. doi: 10.1136/ard.2009.109702. No abstract available. PMID 19822712
- [Background] Lecluse LL, Driessen RJ, Spuls PI, de Jong EM, Stapel SO, van Doorn MB, Bos JD, Wolbink GJ. Extent and clinical consequences of antibody formation against adalimumab in patients with plaque psoriasis. Arch Dermatol. 2010 Feb;146(2):127-32. doi: 10.1001/archdermatol.2009.347. PMID 20157022
- [Background] Ben-Horin S, Yavzori M, Katz L, Kopylov U, Picard O, Fudim E, Coscas D, Bar-Meir S, Goldstein I, Chowers Y. The immunogenic part of infliximab is the F(ab')2, but measuring antibodies to the intact infliximab molecule is more clinically useful. Gut. 2011 Jan;60(1):41-8. doi: 10.1136/gut.2009.201533. Epub 2010 Jun 2. PMID 20519742
- [Background] Karmiris K, Paintaud G, Noman M, Magdelaine-Beuzelin C, Ferrante M, Degenne D, Claes K, Coopman T, Van Schuerbeek N, Van Assche G, Vermeire S, Rutgeerts P. Influence of trough serum levels and immunogenicity on long-term outcome of adalimumab therapy in Crohn's disease. Gastroenterology. 2009 Nov;137(5):1628-40. doi: 10.1053/j.gastro.2009.07.062. Epub 2009 Aug 5. PMID 19664627
- [Background] Nanda KS, Cheifetz AS, Moss AC. Impact of antibodies to infliximab on clinical outcomes and serum infliximab levels in patients with inflammatory bowel disease (IBD): a meta-analysis. Am J Gastroenterol. 2013 Jan;108(1):40-7; quiz 48. doi: 10.1038/ajg.2012.363. Epub 2012 Nov 13. PMID 23147525
- [Background] Vande Casteele N, Gils A, Singh S, Ohrmund L, Hauenstein S, Rutgeerts P, Vermeire S. Antibody response to infliximab and its impact on pharmacokinetics can be transient. Am J Gastroenterol. 2013 Jun;108(6):962-71. doi: 10.1038/ajg.2013.12. Epub 2013 Feb 19. PMID 23419382
- [Background] Steenholdt C, Svenson M, Bendtzen K, Thomsen OO, Brynskov J, Ainsworth MA. Severe infusion reactions to infliximab: aetiology, immunogenicity and risk factors in patients with inflammatory bowel disease. Aliment Pharmacol Ther. 2011 Jul;34(1):51-8. doi: 10.1111/j.1365-2036.2011.04682.x. Epub 2011 May 3. PMID 21535447
- [Background] Afif W, Loftus EV Jr, Faubion WA, Kane SV, Bruining DH, Hanson KA, Sandborn WJ. Clinical utility of measuring infliximab and human anti-chimeric antibody concentrations in patients with inflammatory bowel disease. Am J Gastroenterol. 2010 May;105(5):1133-9. doi: 10.1038/ajg.2010.9. Epub 2010 Feb 9. PMID 20145610
- [Background] Bartelds GM, Krieckaert CL, Nurmohamed MT, van Schouwenburg PA, Lems WF, Twisk JW, Dijkmans BA, Aarden L, Wolbink GJ. Development of antidrug antibodies against adalimumab and association with disease activity and treatment failure during long-term follow-up. JAMA. 2011 Apr 13;305(14):1460-8. doi: 10.1001/jama.2011.406. PMID 21486979
- [Background] Steenholdt C, Brynskov J, Thomsen OO, Munck LK, Fallingborg J, Christensen LA, Pedersen G, Kjeldsen J, Jacobsen BA, Oxholm AS, Kjellberg J, Bendtzen K, Ainsworth MA. Individualised therapy is more cost-effective than dose intensification in patients with Crohn's disease who lose response to anti-TNF treatment: a randomised, controlled trial. Gut. 2014 Jun;63(6):919-27. doi: 10.1136/gutjnl-2013-305279. Epub 2013 Jul 22. PMID 23878167
- [Background] Velayos FS, Kahn JG, Sandborn WJ, Feagan BG. A test-based strategy is more cost effective than empiric dose escalation for patients with Crohn's disease who lose responsiveness to infliximab. Clin Gastroenterol Hepatol. 2013 Jun;11(6):654-66. doi: 10.1016/j.cgh.2012.12.035. Epub 2013 Jan 26. PMID 23357488
- [Background] Paul S, Del Tedesco E, Marotte H, Rinaudo-Gaujous M, Moreau A, Phelip JM, Genin C, Peyrin-Biroulet L, Roblin X. Therapeutic drug monitoring of infliximab and mucosal healing in inflammatory bowel disease: a prospective study. Inflamm Bowel Dis. 2013 Nov;19(12):2568-76. doi: 10.1097/MIB.0b013e3182a77b41. PMID 24013361
- [Background] Roblin X, Marotte H, Rinaudo M, Del Tedesco E, Moreau A, Phelip JM, Genin C, Peyrin-Biroulet L, Paul S. Association between pharmacokinetics of adalimumab and mucosal healing in patients with inflammatory bowel diseases. Clin Gastroenterol Hepatol. 2014 Jan;12(1):80-84.e2. doi: 10.1016/j.cgh.2013.07.010. Epub 2013 Jul 23. PMID 23891927